CLINICAL TRIAL: NCT07103889
Title: Assessment of Biochemical, Metabolic, Inflammatory, and Hematological Parameters Following Acute Exercise in Normal-Weight and Overweight/Obese Adolescent Girls.
Brief Title: Effect of Acute Exercise on Biochemical Parameters in Normal-Weight and Overweight/Obese Adolescent.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: High Institute of Sports and Physical Education of Kef (Other)
Responsible Party: Principal Investigator, Wissal Abassi, Principal Investigator, High Institute of Sports and Physical Education of Kef
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: ACUTE-EXER-OBESE-2025
Record Dates: First submitted 2025-07-18; First posted 2025-08-05 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-07

CONDITIONS: Obese Adolescents; Overweight
Keywords: Adolescent; Maximal Exercise; Blood Biomarkers; Liver Enzymes; Lipid Profile; Renal Function; obesity; overweight; Normal-weight
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Normal-weight adolescent girls (Experimental): Body mass index (BMI) between the 5th and <85th percentile for age.
  Interventions: Behavioral: Spartacus Test
- Overweight/obese adolescent (Experimental): BMI ≥ 85th percentile for age.
  Interventions: Behavioral: Spartacus Test

INTERVENTIONS:
Behavioral: Spartacus Test — The Spartacus test was conducted on a 750 m (75 × 10 m) rectangular course marked with cones at regular intervals to indicate different speeds (from 7 to 18 km/h). Each participant began running at 7 km/h, with speed increasing by 1 km/h every three minutes.During the 3-minute intervals (for each speed stage), participants had 15 seconds to reach the corresponding marker, followed by 15 seconds of rest. Participants had to adjust their running pace to reach the target cone in synchrony with an audio signal. The test ended when a participant failed to reach the next cone within the given time. This test is validated for assessing maximal aerobic capacity (MAS) in obese adolescents. During the Spartacus test, maximal heart rate (HRmax) was recorded using a heart rate monitor (S810; Polar, Kempele, Finland).

SUMMARY:
The goal of this interventional clinical trial is to compare the acute physiological and biochemical responses to maximal physical exercise (Spartacus test). in two groups of adolescent girls: in normal-weight and overweight/obese adolescent. The main question it aims to answer:

* Does Spartacus test significantly alter glucose metabolism and lipid profile in normal-weight and overweight/obese adolescent?
* How do inflammatory markers such as C-Reactive Protein [CRP], Erythrocyte Sedimentation Rate [ESR], respond immediately after and 30 minutes following maximal effort?
* Are there significant changes in liver enzymes (Aspartate Aminotransferase [AST], Alanine Aminotransferase [ALT]), muscle damage indicators (creatine kinase [CK], Lactate Dehydrogenase [LDH]), and electrolyte balance post-exercise? Participants will undergo a baseline blood draw before performing the Spartacus test , a progressive maximal exercise test. Blood samples will then be collected immediately after the test and again 30 minutes post-exercise to evaluate changes in: Glucose metabolism (fasting glucose), Lipid profile (total cholesterol, High-Density Lipoprotein [HDL], Low-Density Lipoprotein [LDL], triglycerides), Liver and muscle enzymes (Aspartate Aminotransferase [AST], Alanine Aminotransferase [ALT], Creatine kinase [CK], Lactate Dehydrogenase [LDH]), Renal function markers (creatinine, urea), Inflammatory markers (C-Reactive Protein [CRP], Erythrocyte Sedimentation Rate [ESR]), Hematological profile (complete blood count: White Blood Cells [WBC], Red Blood Cells [RBC], Hemoglobin [Hb], Hematocrit [Hct], platelets), Electrolytes (sodium, potassium, chloride), Uric acid, calcium, phosphorus, magnesium, iron.

DETAILED DESCRIPTION:
This is an interventional clinical trial designed to evaluate the acute physiological and biochemical responses to maximal physical exercise (Spartacus test) in normal-weight and overweight/obese adolescent. The study aims to investigate how a single session Spartacus test affects key metabolic, inflammatory, hepatic, muscular, renal, and hematological parameters.

Participants will be divided into two groups:

Group 1: Normal-weight adolescent girls Adolescent girls with a body mass index (BMI) between the 5th and <85th percentile for age.

Group 2: Overweight/obese adolescent girls Adolescent girls with a BMI ≥ 85th percentile for age. The protocol involves running on a simulated rectangular course (750 m²), with increasing speed every 3 minutes (starting at 7 km/h and increasing by 1 km/h each stage). Participants must reach a marked cone corresponding to the new speed within 15 seconds, followed by a 15-second rest period before the next stage begins. The test continues until voluntary exhaustion or inability to maintain the required pace.

Blood samples will be collected at three time points:

Baseline (Time 0): Before the start of the exercise. Immediately post-exercise (Time 1): Within 5 minutes after completion of the test.

30 minutes post-exercise (Time 2): To assess early recovery kinetics.

The following biomarkers will be measured at each time point:

Metabolic profile: Fasting glucose, lipid panel (total cholesterol, HDL, LDL, triglycerides), uric acid Liver function: AST, ALT, LDH, CK Renal function: Creatinine, urea Inflammatory markers: C-reactive protein (CRP), erythrocyte sedimentation rate (ESR) Hematological profile: Complete blood count (CBC), including white blood cell differential, hemoglobin, hematocrit, red blood cell indices, and platelet count Electrolytes: Sodium (Na⁺), potassium (K⁺), chloride (Cl-) Minerals and trace elements: Calcium, phosphorus, magnesium, iron

ELIGIBILITY:
Inclusion Criteria:

* Female,
* Aged 14-18 years
* BMI between the 5th and <85th percentile for age (normal-weight group), or BMI ≥ 85th percentile for age (overweight/obese group)
* No chronic illness or contraindication to exercise
* No regular medication use
* Written informed consent from participant and parent/legal guardian

Exclusion Criteria:

* Presence of chronic diseases (diabetes, thyroid disorders, etc.)
* Musculoskeletal or cardiovascular contraindications to maximal exercise
* Pregnancy
* Recent infection or inflammation
* Use of anti-inflammatory or hormonal medications

Ages: 13 Years to 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes — Female
Enrollment: 35 (Actual)
Dates: Start 2025-08-10 (Actual); Primary Completion 2025-08-13 (Actual); Study Completion 2025-08-13 (Actual)

PRIMARY OUTCOMES:
Concentration of Blood Glucose (mg/dL) | At baseline, Immediately after Spartacus, and 30 minutes post-Spartacus.
  Blood glucose levels will be measured using enzymatic colorimetric assays in a certified clinical laboratory.
iron | At baseline, Immediately after Spartacus, and 30 minutes post-Spartacus.
  Serum iron concentration will be measured using a colorimetric assay in a certified clinical laboratory.
Concentration of Total Cholesterol (mg/dL) | At baseline, Immediately after Spartacus, and 30 minutes post-Spartacus.
  Total cholesterol will be assessed using enzymatic colorimetric assays in a certified clinical laboratory.
Concentration of HDL Cholesterol (mg/dL) | At baseline, Immediately after Spartacus, and 30 minutes post-Spartacus.
  HDL cholesterol will be analyzed using enzymatic colorimetric assays in a certified clinical laboratory.
Concentration of Triglycerides (mg/dL) | At baseline, Immediately after Spartacus, and 30 minutes post-Spartacus.
  Triglyceride levels will be measured using enzymatic colorimetric assays in a certified clinical laboratory.
Calculated LDL Cholesterol (mg/dL) | At baseline, Immediately after Spartacus, and 30 minutes post-Spartacus.
  LDL cholesterol will be estimated using the Friedewald formula based on total cholesterol, HDL cholesterol, and triglycerides measured via enzymatic colorimetric assays in a certified clinical laboratory.
  LDL-C (mg/dL)=Cholesterol total-HDL Cholesterol-( Triglycerides /5)
Concentration of C-Reactive Protein (CRP) (mg/L) | At baseline, Immediately after Spartacus, and 30 minutes post-Spartacus.
  CRP levels will be measured using enzymatic colorimetric assays in a certified clinical laboratory.
Erythrocyte Sedimentation Rate (ESR) (mm/hr) | At baseline, Immediately after Spartacus, and 30 minutes post-Spartacus.
  ESR will be determined using standard laboratory methods in a certified clinical laboratory.
Concentration of Aspartate Aminotransferase (AST) (U/L) | At baseline, Immediately after Spartacus, and 30 minutes post-Spartacus.
  AST levels will be measured using enzymatic colorimetric assays in a certified clinical laboratory.
Concentration of Alanine Aminotransferase (ALT) (U/L) | At baseline, Immediately after Spartacus, and 30 minutes post-Spartacus.
  ALT levels will be measured using enzymatic colorimetric assays in a certified clinical laboratory.
Concentration of Lactate Dehydrogenase (LDH) (U/L) | At baseline, Immediately after Spartacus, and 30 minutes post-Spartacus.
  LDH levels will be measured using enzymatic colorimetric assays in a certified clinical laboratory.
Concentration of Creatine Kinase (CK) (U/L) | At baseline, Immediately after Spartacus, and 30 minutes post-Spartacus.
  CK levels will be measured using enzymatic colorimetric assays in a certified clinical laboratory.
Concentration of Creatinine (mg/dL) | At baseline, Immediately after Spartacus, and 30 minutes post-Spartacus.
  Creatinine levels will be measured using enzymatic colorimetric assays in a certified clinical laboratory.
Concentration of Urea (mg/dL) | At baseline, Immediately after Spartacus, and 30 minutes post-Spartacus.
  Urea levels will be measured using enzymatic colorimetric assays in a certified clinical laboratory.
Concentration of Serum Uric Acid (mg/dL) | At baseline, Immediately after Spartacus, and 30 minutes post-Spartacus.
  Serum concentrations of uric acid will be measured using enzymatic colorimetric assays in a certified clinical laboratory.
Glomerular Filtration Rate | At baseline, Immediately after Spartacus, and 30 minutes post-Spartacus.
  The glomerular Filtration Rate (GFR) has been computed using the Cockcroft formula, as follows: GFR (mL/min) = [(140 - age) × weight ×0.85]/( Serum Creatinine× 72).
White Blood Cell Count (WBC) (10³/µL) | At baseline, Immediately after Spartacus, and 30 minutes post-Spartacus.
  WBC will be measured using standard hematology analyzers in a certified clinical laboratory.
Red Blood Cell Count (RBC) (10³/µL) | At baseline, Immediately after Spartacus, and 30 minutes post-Spartacus.
  RBC will be measured using standard hematology analyzers in a certified clinical laboratory.
Hemoglobin Concentration (Hb) (g/dL) | At baseline, Immediately after Spartacus, and 30 minutes post-Spartacus.
  Hb concentration will be measured using standard hematology analyzers in a certified clinical laboratory.
Hematocrit (Hct) (%) | At baseline, Immediately after Spartacus, and 30 minutes post-Spartacus.
  Hematocrit will be measured using standard hematology analyzers in a certified clinical laboratory.
Platelet Count (10³/µL) | At baseline, Immediately after Spartacus, and 30 minutes post-Spartacus.
  Platelet count will be measured using standard hematology analyzers in a certified clinical laboratory.
Mean Corpuscular Hemoglobin Content (MCH) (pg) | At baseline, Immediately after Spartacus, and 30 minutes post-Spartacus.
  Blood levels of mean corpuscular hemoglobin content will be measured from a 5 ml blood sample and analyzed using a multichannel automated hematology analyzer in a certified clinical laboratory.
Mean Hemoglobin Concentration (MCHC) (g/dL) | At baseline, Immediately after Spartacus, and 30 minutes post-Spartacus.
  Blood levels of mean hemoglobin concentration will be measured from a 5 ml blood sample and analyzed using a multichannel automated hematology analyzer in a certified clinical laboratory.
Mean Corpuscular Volume (MCV) (fL) | At baseline, Immediately after Spartacus, and 30 minutes post-Spartacus.
  Blood levels of mean corpuscular volume will be measured from a 5 ml blood sample and analyzed using a multichannel automated hematology analyzer in a certified clinical laboratory
Plasma volume variations | Plasma volume variations (PVV) was calculated Immediately after Spartacus, and 30 minutes post-Spartacus.
  Plasma volume variations (PVV) was calculated based on measured hematocrit (Ht) and hemoglobin (Hb) valuesaccording to the method developed by Costill and Fink (1974). %PVV=100 ×[(HbA/HbB) ×(100 - HtB) / (100 - HtA)] -
  1, where 0 is the value measured before exercise and 1 is the value measured after exercise.
Serum Sodium Concentration (mmol/L) | At baseline, Immediately after Spartacus, and 30 minutes post-Spartacus.
  Serum sodium levels will be measured using enzymatic colorimetric assays in a certified clinical laboratory.
Serum Potassium Concentration (mmol/L) | At baseline, Immediately after Spartacus, and 30 minutes post-Spartacus.
  Serum potassium levels will be measured using enzymatic colorimetric assays in a certified clinical laboratory.
Serum Chloride Concentration (mmol/L) | At baseline, Immediately after Spartacus, and 30 minutes post-Spartacus.
  Serum chloride levels will be measured using enzymatic colorimetric assays in a certified clinical laboratory.
Serum Calcium Concentration (mmol/L) | At baseline, Immediately after Spartacus, and 30 minutes post-Spartacus.
  Serum calcium levels will be measured using enzymatic colorimetric assays in a certified clinical laboratory.
Serum Phosphorus Concentration (mmol/L) | At baseline, Immediately after Spartacus, and 30 minutes post-Spartacus.
  Serum phosphorus levels will be measured using enzymatic colorimetric assays in a certified clinical laboratory.
Serum Magnesium Concentration (mg/dL) | At baseline, Immediately after Spartacus, and 30 minutes post-Spartacus.
  Serum magnesium concentration will be determined using a spectrophotometric colorimetric method in a certified clinical laboratory.
Serum Iron Concentration (µg/dL) | At baseline, Immediately after Spartacus, and 30 minutes post-Spartacus.
  Serum iron concentration will be measured using enzymatic colorimetric assays in a certified clinical laboratory.

CONTACTS AND LOCATIONS:
Overall Officials: Wissal abassi, Dr, Principal Investigator — Research Unit "Sport Sciences, Health and Movement"(UR22JS01) High Institute of Sport and Physical Education of Kef, University of Jendouba, 7100 Kef, Tunisia.
Locations (1):
- High Institute of Sports and Physical Education of Kef, Boulifa, Kef Governorate, Tunisia